CLINICAL TRIAL: NCT01934621
Title: Closing the Gap: Early Intervention for Cognitive Disability After Stroke
Brief Title: Adapting Daily Activity Performance Through Strategy Training
Acronym: ADAPTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Elizabeth R. Skidmore, PhD, OTR/L, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO13070029; R01HD074693 (NIH)
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Strategy Training; Attention Control
Keywords: Stroke; Rehabilitation; Cognition; Disability
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Strategy Training (Experimental): Strategy training is a form of meta-cognitive instruction that trains individuals with stroke-related cognitive impairments to identify and prioritize problematic daily activities, identify the barriers impeding performance, generate and evaluate their own strategies to address barriers, and apply these skills through iterative practice. Participants use printed workbooks to learn and apply this method.
  Interventions: Behavioral: Strategy Training
- Attention Control (Placebo Comparator): The attention control intervention will control for the non-specific effects of strategy training. The therapists will administer the standardized and dose-matched protocol, using scripted open-ended questions to facilitate participants' reflections on their rehabilitation activities and experiences. In lieu of the strategy training workbook materials, participants will complete a daily journal, and discuss their entries during attention control sessions.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Strategy Training
  Arms: Strategy Training
Behavioral: Attention Control
  Arms: Attention Control

SUMMARY:
Individuals with cognitive impairments after stroke sustain significant disability in their daily tasks, and account for a significant proportion of stroke-related healthcare costs. The proposed study examines a novel intervention, strategy training, that shows promise for helping individuals with stroke-related cognitive impairments reduce disability in daily tasks, which may lead to reductions in healthcare costs. We predict that strategy training will result in significantly greater independence 6 months after stroke compared to an attention control intervention, and that strategy training may reduce cognitive impairments.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of acute stroke
* admission to acute inpatient rehabilitation
* impairment in higher order cognitive functions (EXIT-14 ≥ 3)

Exclusion Criteria:

* pre-stroke diagnosis of dementia in the medical record
* inability to follow two- step commands 80% of the time
* severe aphasia (BDAE ≤ 1)
* current major depressive, bipolar, or psychotic disorder
* drug or alcohol abuse within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Change in Independence with Daily Activities | Baseline to Month 6
  Moderate effect size of difference between groups in independence (measured with the Functional Independence Measure)

SECONDARY OUTCOMES:
Change in Executive Functions | Baseline to Month 6
  Moderate effect size of difference between groups in independence (measured with selected indices of the Delis-Kaplan Executive Function System)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R Skidmore, PhD, OTR/L, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Kringle EA, Terhorst L, Butters MA, Skidmore ER. Clinical Predictors of Engagement in Inpatient Rehabilitation Among Stroke Survivors With Cognitive Deficits: An Exploratory Study. J Int Neuropsychol Soc. 2018 Jul;24(6):572-583. doi: 10.1017/S1355617718000085. Epub 2018 Mar 19. PMID 29552996